CLINICAL TRIAL: NCT06463106
Title: Endothelial Dysfunction in Post-infection Fatigue Syndromes
Status: Completed | Type: Observational
Sponsor: FH Joanneum Gesellschaft mbH (Industry)
Responsible Party: Principal Investigator, Francisco Westermeier, PhD, FH Joanneum Gesellschaft mbH
Other Study IDs: FWF_KLP9628023
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Chronic Fatigue Syndrome; Long COVID
Keywords: ME/CFS; Long COVID; Endothelial dysfunction
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Post-infection chronic fatigue syndromes, such as myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) and post-COVID-19 condition (Long Covid), are conditions primarily characterized by debilitating fatigue. This fatigue can range from mild, where patients are still able to participate in some social activities (e.g., school, work), to moderate and severe, where sufferers are predominantly homebound and bedridden. As a result, ME/CFS and Long Covid not only negatively impact the quality of life of affected individuals and their caregivers but also represent a substantial and often silent burden on healthcare systems worldwide, including Austria. This is primarily because most cases remain undiagnosed due to the lack of standardized clinical assessments and diagnostic markers. Endothelial dysfunction, which is well known to affect blood flow, oxygen and nutrient delivery, and waste removal in the body, has been described as one of the key factors behind the symptoms experienced by ME/CFS and Long Covid patients. However, the mechanisms that might explain the development of endothelial dysfunction remain largely unexplored. Therefore, this project aims to evaluate key biological aspects related to the function of endothelial cells - a layer of cells lining blood vessels - using plasma samples from an Austrian cohort of ME/CFS and Long Covid patients. We expect that the findings from our study will provide new insights to better understand endothelial dysfunction in post-infection chronic fatigue syndromes, leading to improved patient stratification and tailored treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for ME/CFS patients not infected with SARS-CoV-2 (n=17; females: 70.59%; age (years): 40.10 ± 10.80) and Long-Covid patients (n=30; females: 73.4%; age (years): 37.70 ± 9.96) include profound fatigue and at least one of the following symptoms: PEM, autonomic dysfunction, and/or orthostatic intolerance. All participants were included only if they were at least 12 weeks past an acute EBV infection and/or 10 weeks past an acute SARS-CoV-2 infection, respectively. SARS-CoV-2 specific IgA (A) and IgG (B) antibody titers were measured using commercial test kits (Anti-SARS-CoV-2-ELISA (IgA) and Anti-SARS-CoV-2-QuantiVac-ELISA (IgG); Euroimmun, Germany) in plasma samples.

Exclusion Criteria:

Participants' exclusion criteria included evidence of acute malignant diseases, diabetes mellitus, acute sepsis, chronic inflammatory gastrointestinal diseases, and frequent intake of analgesics, antacids, or antibiotics. Furthermore, no previously hospitalized SARS-CoV-2 patients were included, eliminating false-positive fatigue due to intensive care treatment, such as artificial respiration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A sex/age-matched cohort (n=107) including (1) healthy controls and patients diagnosed with (2) ME/CFS and (3) Long-Covid according to the ethical approval granted by the Ethics Committee at the Medical University of Vienna (vote number: 2281/2020). Healthy individuals will be divided into two sub-groups: individuals without SARS-CoV-2 infection (HC1; n=30; females: 73.4%; age (years): 34.37 ± 12.30) and previously SARS-CoV-2 infected, fully convalescent patients (HC2; n=30; females: 73.4%; age (years): 34.10 ± 11.51).
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Circulating levels of L-arginine metabolites | 6 months
  Ultra-high performance liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS)
Markers of endothelial inflammation | 6 months
  ELISA
Production of reactive oxygen species (ROS) in endothelial cells | 6 months
  Fluorometric assay
Endothelial permeability | 6 months
  3D culture model
Angiogenesis | 6 months
  3D culture model
Epigenetic and transcriptomic patterns in endothelial cells | 6 months
  Genome wide DNA methylation and RNA sequencing (RNA-seq)

CONTACTS AND LOCATIONS:
Locations (1):
- FH JOANNEUM University of Applied Sciences, Graz, Austria

REFERENCES:
- [Background] Pipper C, Bliem L, Leon LE, Mennickent D, Bodner C, Guzman-Gutierrez E, Stingl M, Untersmayr E, Wagner B, Bertinat R, Sepulveda N, Westermeier F. Sex and disease severity-based analysis of steroid hormones in ME/CFS. J Endocrinol Invest. 2024 Sep;47(9):2235-2248. doi: 10.1007/s40618-024-02334-1. Epub 2024 May 10. PMID 38724880
- [Background] Bertinat R, Villalobos-Labra R, Hofmann L, Blauensteiner J, Sepulveda N, Westermeier F. Decreased NO production in endothelial cells exposed to plasma from ME/CFS patients. Vascul Pharmacol. 2022 Apr;143:106953. doi: 10.1016/j.vph.2022.106953. Epub 2022 Jan 21. PMID 35074481
- [Background] Blauensteiner J, Bertinat R, Leon LE, Riederer M, Sepulveda N, Westermeier F. Altered endothelial dysfunction-related miRs in plasma from ME/CFS patients. Sci Rep. 2021 May 19;11(1):10604. doi: 10.1038/s41598-021-89834-9. PMID 34011981
- See also: FWF / Austrian Science Fund — http://www.fwf.ac.at/forschungsradar/10.55776/KLP9628023